CLINICAL TRIAL: NCT06372145
Title: An Interventional, Phase 3 Extension Study to Investigate Long-term Safety and Tolerability of Tolebrutinib in Participants With Relapsing Multiple Sclerosis, Primary Progressive Multiple Sclerosis, or Nonrelapsing Secondary Progressive Multiple Sclerosis
Brief Title: A Study to Investigate Long-term Safety and Tolerability of Tolebrutinib in Participants With Multiple Sclerosis.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTS17043; 2023-503631-18 (Registry Identifier: CTIS); U1111-1287-6797 (Registry Identifier: ICTRP)
Record Dates: First submitted 2024-04-15; First posted 2024-04-17 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Relapsing Multiple Sclerosis; Secondary Progressive Multiple Sclerosis; Progressive Relapsing Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive | interventions — teriflunomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tolebrutinib (Experimental): * Participants will receive OL tolebrunitib 60 mg once daily.
  * RMS participants who are not eligible for OL tolebrutinib per Health Authority and/or ethics committee decisions on the study conduct (ie, partial hold on initiation of tolebrutinib) will continue their parent study treatment assignment as per their randomization from the parent study.
  Interventions: Drug: Tolebrutinib; Drug: Placebo
- Teriflunomide (Active Comparator): * participants will receive teriflunomide 14 mg daily
  * RMS participants who are not eligible for OL tolebrutinib per Health Authority and/or ethics committee decisions on the study conduct (ie, partial hold on initiation of tolebrutinib) will continue their parent study treatment assignment (either tolebrutinib or teriflunomide) as per their randomization from the parent study. If unblinded to teriflunomide parent study treatment assignment, these RMS participants will continue teriflunomide in the LTS17043 study.
  Interventions: Drug: Placebo; Drug: Teriflunomide

INTERVENTIONS:
Drug: Tolebrutinib — Pharmaceutical form:Tablet-Route of administration:oral
  Other Names: SAR442168
  Arms: Tolebrutinib
Drug: Placebo — Pharmaceutical form:Tablet-Route of administration:oral
Drug: Teriflunomide — Pharmaceutical form:Tablet-Route of administration:oral
  Other Names: Aubagio
  Arms: Teriflunomide

SUMMARY:
This is a Phase 3 extension, global, multicenter study to assess the long-term safety and tolerability of tolebrutinib in adult participants (aged ≥18 years) with RMS, PPMS, or NRSPMS who were previously enrolled in the Phase 2b LTS (LTS16004) or 1 of the 4 Phase 3 tolebrutinib pivotal trials (GEMINI 1 [EFC16033], GEMINI 2 [EFC16034], HERCULES [EFC16645], or PERSEUS [EFC16035]).

SUBSTUDY: ToleDYNAMIC substudy

DETAILED DESCRIPTION:
Participants with relapsing MS from the Phase 2b LTS16004 parent study will continue open-label (OL) tolebrutinib.

All participants from the Phase 3 parent studies (EFC16033, EFC16034, EFC16645, and EFC16035) will learn which treatment they received in the parent study:

* If from one of the Phase 3 relapsing MS studies and on teriflunomide, an accelerated elimination procedure or a 3-month washout period is required prior to starting OL tolebrutinib. If on teriflunomide, and benefiting and recommended by the Investigator, the participant may opt to continue teriflunomide outside of the LTS17043 study, if clinically appropriate. If on tolebrutinib, the participant will continue tolebrutinib.
* All participants from one of the Phase 3 progressive MS studies will start OL tolebrutinib.
* If a participant already started OL tolebrutinib in the Phase 3 parent study this will be continued.
* RMS participants who are not eligible for OL tolebrutinib per Health Authority and/or ethics committee decisions on the study conduct (ie, partial hold on initiation of tolebrutinib) will continue their parent study treatment assignment as per their randomization from the parent study.

The treatment duration per participant will be approximately 3 years of OL tolebrutinib.

ELIGIBILITY:
Inclusion Criteria:

- Participants with RMS, PPMS, or NRSPMS who completed the Phase 2b LTS (LTS16004) or 1 of the 4 Phase 3 pivotal tolebrutinib trials (EFC16033, EFC16034, EFC16645, EFC16035) on IMP.

OR

- The Phase 2b LTS (LTS16004) or Phase 3 tolebrutinib pivotal trial participants who temporarily discontinued IMP due to a national emergency and completed the trial visits.

ToleDYNAMIC Substudy: Inclusion criteria are those of the main study

Exclusion Criteria:

* Participants are excluded from the study if any of the following criteria apply:
* The participant is at risk for or has a persistent chronic, active (including fever higher than 38°C and clinically unstable), or recurring systemic infection, as judged by the Investigator
* For participants initiating OL tolebrutinib in the LTS17043 study: Participants at risk of developing or having reactivation of hepatitis, ie, results at the unblinding visit (RMS) or opt-in visit (PMS) for serological markers for hepatitis B and C viruses indicating acute or chronic infection
* Active alcohol use disorder or a history of alcohol or drug abuse within 1 year prior to the opt-in visit
* Current alcohol intake equal to or exceeding the following at the opt-in visit: more than 2 drinks per day for men and more than 1 drink per day for women
* Abnormal ECG during the opt-in visit considered in the Investigator's judgment to be clinically significant, such as QTcF >500 msec, in the context of this study.
* A bleeding disorder, known platelet dysfunction, abnormal platelet count (<100,000/microliter), history of significant bleeding event or other conditions and planned procedures that may predispose the participant to excessive bleeding during the study, as judged by the Investigator.
* For participants initiating OL tolebrutinib in the LTS17043 study: Confirmed unblinding visit (RMS) or opt-in visit (PMS) alanine aminotransferase (ALT) more than 1.5 × upper limit of normal (ULN) OR aspartate aminotransferase (AST) more than 1.5 × ULN OR alkaline phosphatase more than 2 × ULN (unless caused by non-liver-related disorder or explained by a stable chronic liver disorder) OR total bilirubin more than 1.5 × ULN (unless due to Gilbert syndrome or non-liver-related disorder).
* Acute liver disease, cirrhosis, chronic liver disease (unless considered stable for more than 6 months).
* Participants who developed clinically relevant cardiovascular, hepatic, endocrine, neuropsychiatric or other major systemic disease making implementation of the protocol or interpretation of the trial results difficult or that would put the patient at risk by participating in the trial, as judged by the Investigator.
* The participant is receiving treatment during the study period with drugs not permitted by the study protocol, including potent and moderate inducers of cytochrome P450 (CYP) 3A or potent inhibitors of CYP2C8 hepatic enzymes.

NOTE: The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

ToleDYNAMIC Substudy: Exclusion criteria are those of the main study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs), Adverse Events of Special Interest (AESIs) and AEs leading to permanent study intervention discontinuation | From baseline until the End of study approximately 3 years per participant
Number of Participants with Potentially clinically significant abnormalities (PCSAs) | From baseline until the End of study approximately 3 years per participant
  Potentially clinically significant abnormalities (PCSAs) determined by laboratory tests, electrocardiogram (ECG), or vital signs and safety findings on MRI during the study period.

SECONDARY OUTCOMES:
Time to onset of 6-month confirmed disability worsening (CDW for RMS) or confirmed disability progression (CDP for PPMS and NRSPMS) for participants from pivotal studies | From baseline until the End of study approximately 3 years per participant
  Time to onset is defined as a sustained increase from baseline EDSS (pivotal trial) of:
  * RMS: ≥1.5 points when the baseline score is 0, ≥1.0 point when the baseline score is 0.5 to ≤5.5 or ≥0.5 point when the baseline score is >5.5
  * PPMS: ≥1.0 point when the baseline score is ≤5.5 or ≥0.5 point when the baseline score is >5.5
  * NRSPMS: ≥1.0 point when the baseline score is ≤5.0 or ≥0.5 point when the baseline score is >5.0
Annualized Relapse Rate (ARR) for RMS only | From baseline until the End of study approximately 3 years per participant
  ARR during the OL treatment period assessed by confirmed protocol-defined relapses
Number of new and/or enlarging T2-hyperintense lesions per year | From baseline until the End of study approximately 3 years per participant
Change from baseline in total volume of T2-hyperintense lesions | From baseline until the End of study approximately 3 years per participant
ToleDYNAMIC substudy Change from baseline in biomarkers | From baseline until 12 months per participant

CONTACTS AND LOCATIONS:
Locations (353):
- United States (52):
  - University of Alabama at Birmingham- Site Number : 8400013, Birmingham, Alabama
  - North Central Neurology Associates- Site Number : 8400009, Cullman, Alabama
  - Center for Neurology and Spine - Phoenix - North 32nd Street- Site Number : 8400089, Phoenix, Arizona
  - UCSD - Altman Clinical and Translational Research Institute (ACTRI)- Site Number : 8400101, La Jolla, California
  - Collaborative Neuroscience Research- Site Number : 8400045, Los Alamitos, California
  - Keck School of Medicine of University of Southern California- Site Number : 8400143, Los Angeles, California
  - Private Practice - Dr. Regina Berkovich- Site Number : 8400059, West Hollywood, California
  - University of Colorado - Anschutz Medical Campus- Site Number : 8400012, Aurora, Colorado
  - Advanced Neurology of Colorado- Site Number : 8400025, Fort Collins, Colorado
  - MedStar Georgetown University Hospital- Site Number : 8400119, Washington D.C., District of Columbia
  - SFM Clinical Research- Site Number : 8400029, Boca Raton, Florida
  - Norman Fixel Institute for Neurological Diseases (FIND)- Site Number : 8400159, Gainesville, Florida
  - Neurology Associates - Maitland- Site Number : 8409902, Maitland, Florida
  - University of Miami Hospital- Site Number : 8400063, Miami, Florida
  - Aqualane Clinical Research- Site Number : 8400027, Naples, Florida
  - Axiom Clinical Research of Florida- Site Number : 8400001, Tampa, Florida
  - University of South Florida- Site Number : 8409905, Tampa, Florida
  - Velocity Clinical Research - Savannah Neurology- Site Number : 8409903, Savannah, Georgia
  - Consultants in Neurology- Site Number : 8409906, Northbrook, Illinois
  - Springfield Clinic 1st - 900 Building- Site Number : 8400071, Springfield, Illinois
  - IU Health Physicians - Fort Wayne - Hope Drive- Site Number : 8400039, Fort Wayne, Indiana
  - University of Kansas Medical Center- Site Number : 8400023, Kansas City, Kansas
  - University of Kentucky Chandler Medical Center- Site Number : 8400106, Lexington, Kentucky
  - Norton Neurology Services- Site Number : 8400127, Louisville, Kentucky
  - The NeuroMedical Center- Site Number : 8400057, Baton Rouge, Louisiana
  - Ochsner Medical Center - Jefferson Highway- Site Number : 8400107, New Orleans, Louisiana
  - Tufts Medical Center- Site Number : 8400072, Boston, Massachusetts
  - UMass Memorial Medical Center - University Campus- Site Number : 8400014, Worcester, Massachusetts
  - Harper University Hospital- Site Number : 8400046, Detroit, Michigan
  - Michigan Institute for Neurological Disorders- Site Number : 8400058, Farmington Hills, Michigan
  - Memorial Healthcare Institute for Neuroscience- Site Number : 8400033, Owosso, Michigan
  - Minneapolis Clinic of Neurology - Golden Valley- Site Number : 8400051, Golden Valley, Minnesota
  - Mayo Clinic in Rochester - Minnesota- Site Number : 8400111, Rochester, Minnesota
  - Sharlin Health and Neurology- Site Number : 8400093, Ozark, Missouri
  - Missouri Baptist Medical Center- Site Number : 8400019, St Louis, Missouri
  - Cleveland Clinic Lou Ruvo Center for Brain Health Las Vegas- Site Number : 8400117, Las Vegas, Nevada
  - The University of New Mexico- Site Number : 8400032, Albuquerque, New Mexico
  - The Mount Sinai Hospital- Site Number : 8400038, New York, New York
  - South Shore Neurologic Associates - Patchogue- Site Number : 8400100, Patchogue, New York
  - Stony Brook University- Site Number : 8400042, Stony Brook, New York
  - Atrium Health - Wake Forest Baptist Medical Center- Site Number : 8400116, Winston-Salem, North Carolina
  - Dayton Center for Neurological Disorders- Site Number : 8400081, Centerville, Ohio
  - Cleveland Clinic - Cleveland- Site Number : 8400125, Cleveland, Ohio
  - The Ohio State University- Site Number : 8400150, Columbus, Ohio
  - The Boster Center for Multiple Sclerosis- Site Number : 8400147, Columbus, Ohio
  - UC Health - Elizabeth Place- Site Number : 8409901, Dayton, Ohio
  - Providence St. Vincent's Medical Center- Site Number : 8400020, Portland, Oregon
  - Premier Neurology- Site Number : 8400069, Greer, South Carolina
  - Hope Neurology- Site Number : 8409904, Knoxville, Tennessee
  - Neurology Center of San Antonio- Site Number : 8400036, San Antonio, Texas
  - University of Vermont Medical Center- Site Number : 8400130, Burlington, Vermont
  - Neurological Associates - Richmond- Site Number : 8400097, Richmond, Virginia
- Argentina (9):
  - Investigational Site Number : 0320003, Rosario, Santa Fe Province
  - Investigational Site Number : 0320005, San Miguel de Tucumán, Tucumán Province
  - Investigational Site Number : 0320002, Buenos Aires
  - Investigational Site Number : 0320004, Buenos Aires
  - Investigational Site Number : 0320007, Buenos Aires
  - Investigational Site Number : 0320001, Buenos Aires
  - Investigational Site Number : 0329901, Buenos Aires
  - Investigational Site Number : 0320006, Córdoba
  - Investigational Site Number : 0320005, San Miguel de Tucumán
- Australia (3):
  - Investigational Site Number : 0360001, Saint Leonards, New South Wales
  - Investigational Site Number : 0360006, Kent Town, South Australia
  - Investigational Site Number : 0360007, Melbourne, Victoria
- Austria (3):
  - Investigational Site Number : 0400003, Innsbruck
  - Investigational Site Number : 0400004, Linz
  - Investigational Site Number : 0400002, Vienna
- Belgium (7):
  - Investigational Site Number : 0560005, Bruges
  - Investigational Site Number : 0560009, Brussels
  - Investigational Site Number : 0560007, Brussels
  - Investigational Site Number : 0560004, Ghent
  - Investigational Site Number : 0560006, Leuven
  - Investigational Site Number : 0560008, Liège
  - Investigational Site Number : 0560001, Overpelt
- Brazil (4):
  - Universidade Federal de Goias- Site Number : 0760003, Goiânia, Goiás
  - Instituto de Neurologia de Curitiba - Ecoville- Site Number : 0760002, Curitiba, Paraná
  - Hospital São Lucas da PUCRS - Porto Alegre - Avenida Ipiranga- Site Number : 0760001, Porto Alegre, Rio Grande do Sul
  - CPHosp Medicina, Ensino e Pesquisa (CPQuali)- Site Number : 0760007, São Paulo
- Bulgaria (8):
  - Investigational Site Number : 1000002, Pleven
  - Investigational Site Number : 1000005, Plovdiv
  - Investigational Site Number : 1000004, Sofia
  - Investigational Site Number : 1000008, Sofia
  - Investigational Site Number : 1000001, Sofia
  - Investigational Site Number : 1000006, Sofia
  - Investigational Site Number : 1000011, Sofia
  - Investigational Site Number : 1000009, Sofia
- Canada (14):
  - Investigational Site Number : 1240002, Edmonton, Alberta
  - Investigational Site Number : 1240017, Burnaby, British Columbia
  - Investigational Site Number : 1249901, Vancouver, British Columbia
  - Investigational Site Number : 1240011, Halifax, Nova Scotia
  - Investigational Site Number : 1240012, Hamilton, Ontario
  - Investigational Site Number : 1240003, Ottawa, Ontario
  - Investigational Site Number : 1240008, Toronto, Ontario
  - Investigational Site Number : 1240013, Toronto, Ontario
  - Investigational Site Number : 1240006, Gatineau, Quebec
  - Investigational Site Number : 1240021, Lévis, Quebec
  - Investigational Site Number : 1240004, Montreal, Quebec
  - Investigational Site Number : 1240015, Montreal, Quebec
  - Investigational Site Number : 1240001, Québec, Quebec
  - Investigational Site Number : 1240007, Sherbrooke, Quebec
- Chile (4):
  - Investigational Site Number : 1520002, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520005, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520001, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520003, Santiago
- China (21):
  - Investigational Site Number : 1560009, Beijing
  - Investigational Site Number : 1560006, Beijing
  - Investigational Site Number : 1560023, Beijing
  - Investigational Site Number : 1560025, Beijing
  - Investigational Site Number : 1560004, Changchun
  - Investigational Site Number : 1560015, Changsha
  - Investigational Site Number : 1560005, Chengdu
  - Investigational Site Number : 1560019, Chongqing
  - Investigational Site Number : 1560035, Fuzhou
  - Investigational Site Number : 1569903, Guangzhou
  - Investigational Site Number : 1560027, Hohhot
  - Investigational Site Number : 1560014, Jiazhuang
  - Investigational Site Number : 1560044, Nanjing
  - Investigational Site Number : 1560042, Nanjing
  - Investigational Site Number : 1569901, Shanghai
  - Investigational Site Number : 1560018, Shenyang
  - Investigational Site Number : 1560008, Taiyuan
  - Investigational Site Number : 1560020, Tianjin
  - Investigational Site Number : 1560026, Wenzhou
  - Investigational Site Number : 1560011, Wuhan
  - Investigational Site Number : 1560017, Xi'an
- Investigational Site Number : 1700001, Bogotá, Colombia
- Croatia (2):
  - Investigational Site Number : 1910001, Zagreb
  - Investigational Site Number : 1910002, Zagreb
- Czechia (11):
  - Investigational Site Number : 2039907, Brno
  - Investigational Site Number : 2030002, Brno
  - Investigational Site Number : 2039903, Hradec Králové
  - Investigational Site Number : 2039901, Jihlava
  - Investigational Site Number : 2039902, Ostrava
  - Investigational Site Number : 2039904, Pardubice
  - Investigational Site Number : 2030008, Prague
  - Investigational Site Number : 2039906, Prague
  - Investigational Site Number : 2039905, Prague
  - Investigational Site Number : 2030003, Teplice
  - Investigational Site Number : 2030007, Zlín
- Denmark (3):
  - Investigational Site Number : 2080001, Esbjerg
  - Investigational Site Number : 2080005, Holstebro
  - Investigational Site Number : 2080004, Odense
- Investigational Site Number : 2330001, Tallinn, Estonia
- Finland (2):
  - Investigational Site Number : 2460001, Tampere
  - Investigational Site Number : 2460002, Turku
- France (16):
  - Investigational Site Number : 2500019, Besançon
  - Investigational Site Number : 2500011, Bron
  - Investigational Site Number : 2500005, Clermont-Ferrand
  - Investigational Site Number : 2500015, Gonesse
  - Investigational Site Number : 2500009, Lille
  - Investigational Site Number : 2500006, Montpellier
  - Investigational Site Number : 2500008, Nancy
  - Investigational Site Number : 2500002, Nice
  - Investigational Site Number : 2500017, Nîmes
  - Investigational Site Number : 2500007, Paris
  - Investigational Site Number : 2500014, Paris
  - Investigational Site Number : 2500004, Poissy
  - Investigational Site Number : 2500003, Rennes
  - Investigational Site Number : 2500010, Saint-Herblain
  - Investigational Site Number : 2500001, Strasbourg
  - Investigational Site Number : 2500012, Toulouse
- Georgia (3):
  - Investigational Site Number : 2680009, Tbilisi
  - Investigational Site Number : 2680003, Tbilisi
  - Investigational Site Number : 2680004, Tbilisi
- Germany (14):
  - Investigational Site Number : 2760005, Bayreuth
  - Investigational Site Number : 2760009, Berlin
  - Investigational Site Number : 2760015, Berlin
  - Investigational Site Number : 2760014, Berlin
  - Investigational Site Number : 2760020, Bochum
  - Investigational Site Number : 2760001, Dresden
  - Investigational Site Number : 2769901, Düsseldorf
  - Investigational Site Number : 2760012, Essen
  - Investigational Site Number : 2760002, Giessen
  - Investigational Site Number : 2760016, Hamburg
  - Investigational Site Number : 2760018, Munich
  - Investigational Site Number : 2760008, Münster
  - Investigational Site Number : 2760011, Ulm
  - Investigational Site Number : 2760003, Würzburg
- Greece (7):
  - Investigational Site Number : 3000006, Athens
  - Investigational Site Number : 3000001, Athens
  - Investigational Site Number : 3000002, Athens
  - Investigational Site Number : 3000007, Athens
  - Investigational Site Number : 3000004, Larissa
  - Investigational Site Number : 3000003, Thessaloniki
  - Investigational Site Number : 3000009, Thessaloniki
- Investigational Site Number : 3440001, Shatin, Hong Kong
- Hungary (4):
  - Investigational Site Number : 3489901, Budapest
  - Investigational Site Number : 3480007, Budapest
  - Investigational Site Number : 3489903, Budapest
  - Investigational Site Number : 3480002, Pécs
- India (9):
  - Investigational Site Number : 3560014, Bengaluru
  - Investigational Site Number : 3569904, Chandigarh
  - Investigational Site Number : 3560007, Gurugram
  - Investigational Site Number : 3569903, Gurugram
  - Investigational Site Number : 3569901, Mangaluru
  - Investigational Site Number : 3560009, Nagpur
  - Investigational Site Number : 3569902, New Delhi
  - Investigational Site Number : 3560002, New Delhi
  - Investigational Site Number : 3560004, Thiruvananthapuram
- Israel (4):
  - Investigational Site Number : 3760003, Haifa
  - Investigational Site Number : 3760001, Ramat Gan
  - Investigational Site Number : 3760006, Rehovot
  - Investigational Site Number : 3760004, Safed
- Italy (16):
  - Investigational Site Number : 3800012, Florence, Firenze
  - Investigational Site Number : 3800016, Florence, Firenze
  - Investigational Site Number : 3800014, Genoa, Genova
  - Investigational Site Number : 3800002, Pozzilli, Isernia
  - Investigational Site Number : 3800001, Milan, Milano
  - Investigational Site Number : 3800010, Milan, Milano
  - Investigational Site Number : 3800006, Naples, Napoli
  - Investigational Site Number : 3800005, Rome, Roma
  - Investigational Site Number : 3800009, Rome, Roma
  - Investigational Site Number : 3800013, Rome, Roma
  - Investigational Site Number : 3800011, Bergamo
  - Investigational Site Number : 3800007, Cagliari
  - Investigational Site Number : 3800015, Catania
  - Investigational Site Number : 3800018, Chieti
  - Investigational Site Number : 3800008, Pavia
  - Investigational Site Number : 3800009, Roma
- Japan (11):
  - Investigational Site Number : 3920022, Morioka, Iwate
  - Investigational Site Number : 3920023, Sagamihara, Kanagawa
  - Investigational Site Number : 3920020, Sendai, Miyagi
  - Investigational Site Number : 3920001, Osaka, Osaka
  - Investigational Site Number : 3920018, Kawagoe, Saitama
  - Investigational Site Number : 3920016, Chiba
  - Investigational Site Number : 3920011, Kyoto
  - Investigational Site Number : 3920004, Osaka
  - Investigational Site Number : 3920014, Tokyo
  - Investigational Site Number : 3920010, Tokyo
  - Investigational Site Number : 3920015, Toyama
- Latvia (2):
  - Investigational Site Number : 4280002, Riga
  - Investigational Site Number : 4280003, Riga
- Lithuania (3):
  - Investigational Site Number : 4400003, Kaunas
  - Investigational Site Number : 4400004, Šiauliai
  - Investigational Site Number : 4400001, Vilnius
- Mexico (4):
  - Investigational Site Number : 4840004, Guadalajara, Jalisco
  - Investigational Site Number : 4840002, Mexico City, Mexico City
  - Investigational Site Number : 4840001, Mexico City, Mexico City
  - Investigational Site Number : 4840003, Veracruz
- Netherlands (4):
  - Investigational Site Number : 5280001, Amsterdam
  - Investigational Site Number : 5280003, Breda
  - Investigational Site Number : 5280006, Groningen
  - Investigational Site Number : 5280002, Heerlen
- Norway (2):
  - Investigational Site Number : 5780003, Bergen
  - Investigational Site Number : 5780001, Oslo
- Poland (10):
  - Investigational Site Number : 6160008, Plewiska, Greater Poland Voivodeship
  - Investigational Site Number : 6160003, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Investigational Site Number : 6160012, Lublin, Lublin Voivodeship
  - Investigational Site Number : 6160001, Lodz, Lódzkie
  - Investigational Site Number : 6160005, Warsaw, Masovian Voivodeship
  - Investigational Site Number : 6160006, Warsaw, Masovian Voivodeship
  - Investigational Site Number : 6160009, Głogów Małopolski, Podkarpackie Voivodeship
  - Investigational Site Number : 6160004, Katowice, Silesian Voivodeship
  - Investigational Site Number : 6160002, Katowice, Silesian Voivodeship
  - Investigational Site Number : 6160011, Zabrze, Silesian Voivodeship
- Portugal (8):
  - Investigational Site Number : 6200001, Braga
  - Investigational Site Number : 6200005, Coimbra
  - Investigational Site Number : 6200011, Lisbon
  - Investigational Site Number : 6200007, Lisbon
  - Investigational Site Number : 6200012, Lisbon
  - Investigational Site Number : 6200006, Lisbon
  - Investigational Site Number : 6200002, Matosinhos Municipality
  - Investigational Site Number : 6200004, Santa Maria da Feira
- San Juan MS Center- Site Number : 8400015, Guaynabo, Puerto Rico
- Romania (8):
  - Investigational Site Number : 6420015, Brasov
  - Investigational Site Number : 6420008, Bucharest
  - Investigational Site Number : 6420004, Campulung Muscel
  - Investigational Site Number : 6420006, Cluj-Napoca
  - Investigational Site Number : 6420003, Constanța
  - Investigational Site Number : 6420013, Oradea
  - Investigational Site Number : 6420005, Sibiu
  - Investigational Site Number : 6420002, Timișoara
- Serbia (5):
  - Investigational Site Number : 6880001, Belgrade
  - Investigational Site Number : 6880003, Belgrade
  - Investigational Site Number : 6880006, Belgrade
  - Investigational Site Number : 6880002, Kragujevac
  - Investigational Site Number : 6880005, Novi Sad
- Slovakia (3):
  - Investigational Site Number : 7030001, Bratislava
  - Investigational Site Number : 7030002, Martin
  - Investigational Site Number : 7030004, Nitra
- Investigational Site Number : 7100001, Pretoria, South Africa
- South Korea (4):
  - Investigational Site Number : 4100001, Goyang-si, Gyeonggi-do
  - Investigational Site Number : 4100003, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100006, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100002, Seoul, Seoul-teukbyeolsi
- Spain (21):
  - Investigational Site Number : 7249908, A Coruña, A Coruña [La Coruña]
  - Investigational Site Number : 7249921, Santiago de Compostela, A Coruña [La Coruña]
  - Investigational Site Number : 7249916, Murcia, Almería
  - Investigational Site Number : 7249906, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7249913, Barakaldo, Basque Country
  - Investigational Site Number : 7249912, Barcelona, Catalunya [Cataluña]
  - Investigational Site Number : 7249919, L'Hospitalet de Llobregat, Catalunya [Cataluña]
  - Investigational Site Number : 7249918, Donostia / San Sebastian, Gipuzkoa
  - Investigational Site Number : 7249911, Girona, Girona [Gerona]
  - Investigational Site Number : 7249904, Las Palmas de Gran Canaria, Las Palmas
  - Investigational Site Number : 7249902, Lleida, Lleida [Lérida]
  - Investigational Site Number : 7249901, Majadahonda, Madrid
  - Investigational Site Number : 7249905, Pozuelo de Alarcón, Madrid
  - Investigational Site Number : 7249907, Seville, Sevilla
  - Investigational Site Number : 7249914, Córdoba
  - Investigational Site Number : 7249909, Madrid
  - Investigational Site Number : 7249903, Madrid
  - Investigational Site Number : 7249910, Madrid
  - Investigational Site Number : 7249915, Málaga
  - Investigational Site Number : 7249920, Palma
  - Investigational Site Number : 7249917, Valencia
- Sweden (2):
  - Investigational Site Number : 7520001, Gothenburg
  - Investigational Site Number : 7520002, Stockholm
- Investigational Site Number : 7560002, Bern, Switzerland
- Taiwan (2):
  - Investigational Site Number : 1580007, Hsinchu
  - Investigational Site Number : 1580002, Taipei
- Investigational Site Number : 7640001, Bangkok, Thailand
- Turkey (Türkiye) (13):
  - Investigational Site Number : 7920006, Ankara
  - Investigational Site Number : 7920005, Eskişehir
  - Investigational Site Number : 7920002, Istanbul
  - Investigational Site Number : 7920009, Istanbul
  - Investigational Site Number : 7920007, Istanbul
  - Investigational Site Number : 7920003, Istanbul
  - Investigational Site Number : 7920014, Izmir
  - Investigational Site Number : 7920010, Izmir
  - Investigational Site Number : 7920001, İzmit
  - Investigational Site Number : 7920017, Konya
  - Investigational Site Number : 7929901, Kütahya
  - Investigational Site Number : 7929902, Mersin
  - Investigational Site Number : 7929903, Samsun
- Ukraine (17):
  - Investigational Site Number : 8040020, Chernivtsi
  - Investigational Site Number : 8049912, Chernivtsi
  - Investigational Site Number : 8049904, Chernivtsi
  - Investigational Site Number : 8049905, Dnipro
  - Investigational Site Number : 8049908, Ivano-Frankivsk
  - Investigational Site Number : 8040025, Kharkiv
  - Investigational Site Number : 8049903, Kharkiv
  - Investigational Site Number : 8040018, Kharkiv
  - Investigational Site Number : 8049902, Kyiv
  - Investigational Site Number : 8049911, Kyiv
  - Investigational Site Number : 8049901, Kyiv
  - Investigational Site Number : 8049914, Lutsk
  - Investigational Site Number : 8049909, Lviv
  - Investigational Site Number : 8049906, Lviv
  - Investigational Site Number : 8049913, Odesa
  - Investigational Site Number : 8049910, Vinnytsia
  - Investigational Site Number : 8040024, Vinnytsia
- United Kingdom (11):
  - Investigational Site Number : 8260009, Bristol, Bristol, City of
  - Investigational Site Number : 8260001, Cardiff, Cardiff [Caerdydd Gb-crd]
  - Investigational Site Number : 8260003, Exeter, Devon
  - Investigational Site Number : 8260005, London, England
  - Investigational Site Number : 8260014, Newcastle upon Tyne, England
  - Investigational Site Number : 8260016, Canterbury, Kent
  - Investigational Site Number : 8260006, London, London, City of
  - Investigational Site Number : 8260019, Salford, Manchester
  - Investigational Site Number : 8260012, Nottingham, Nottinghamshire
  - Investigational Site Number : 8260013, Oxford, Oxfordshire
  - Investigational Site Number : 8260010, Swansea, Swansea [Abertawe Gb-ata]

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: LTS17043 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25716&tenant=MT_SNY_9011